CLINICAL TRIAL: NCT00093665
Title: A Phase II Study Of Alternating Chemoradiotherapy For Nasopharyngeal Cancer Using Cisplatin And 5-Fluorouracil
Brief Title: Fluorouracil, Cisplatin, and Radiation Therapy in Treating Patients With Stage II, Stage III, or Stage IV Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aichi Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: AICHI-UHA-HN03-01; CDR0000389425 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2006-10

CONDITIONS: Head and Neck Cancer
Keywords: stage II lymphoepithelioma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Fluorouracil; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining fluorouracil and cisplatin with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving fluorouracil and cisplatin together with radiation therapy works in treating patients with stage II, stage III, or stage IV nasopharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine progression-free survival of patients with previously untreated stage IIB-IVB nasopharyngeal cancer treated with fluorouracil, cisplatin, and radiotherapy.

Secondary

* Determine overall survival and response rate in patients treated with this regimen.
* Determine compliance to this regimen in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive chemotherapy comprising fluorouracil IV continuously on days 1-5 and cisplatin IV continuously on days 6-7. Beginning 2-3 days after the completion of chemotherapy, patients undergo radiotherapy once daily, 5 days a week, for 4 weeks. With 2-3 days between each course, patients receive a second course of chemotherapy, undergo a second course of radiotherapy, and then receive a third course of chemotherapy. Treatment continues in the absence of unacceptable toxicity or disease progression.

Patients are followed for 3 years.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nasopharyngeal cancer (NPC)

  * Type I-III disease by WHO classification
  * Stage IIB-IVB disease by TNM classification with no distant metastases by chest x-ray, liver ultrasonography or CT scan, and bone scintigraphy

    * Lymph node metastases evaluated by CT scan, MRI, and palpation
  * Progression range of primary lesion evaluated by MRI and pharyngeal fiberoptic endoscopy

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* No severe hepatic dysfunction

Renal

* Creatinine clearance > 60 mL/min
* No severe renal dysfunction

Cardiovascular

* No severe cardiac dysfunction

Pulmonary

* No severe pulmonary dysfunction

Other

* No other active cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for NPC

Chemotherapy

* No prior systemic chemotherapy for NPC

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2003-11

PRIMARY OUTCOMES:
Progression-free survival at 3 years

SECONDARY OUTCOMES:
Overall survival
Response rate
Treatment completion rate
Incidence of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Nobukazu Fuwa, Study Chair — Aichi Cancer Center
Locations (7):
- Japan (7):
  - National Hospital Organization - Medical Center of Kure, Hiroshima
  - Kanazawa University, Kanazawa
  - Kyoto Prefectural University of Medicine, Kyoto
  - Aichi Cancer Center, Nagoya
  - Nara Medical University Cancer Center, Nara
  - Graduate School of Medical Science at the University of Ryukyu, Okinawa
  - Mie University School of Medicine, Tsu